CLINICAL TRIAL: NCT01477190
Title: Spinal Analgesia for Colonic Resection Using an Enhanced Recovery After Surgery (ERAS) Program
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriele Baldini, Assistant Professor, Dr, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN-06-023(2)
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Colon Cancer; Inflammatory Bowel Diseases; Diverticulitis
MeSH Terms: conditions — Colonic Neoplasms; Inflammatory Bowel Diseases; Diverticulitis | interventions — Anesthesia, Spinal; Passive Cutaneous Anaphylaxis; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal group (Experimental): Isobaric bupivacaine 0.5% 10 mg together with preservative-free morphine was injected. The dose of morphine was based on patient's age, with 200 μg in patients aged ≤ 75 years and 150 μg in patients aged > 75 years.
  Interventions: Drug: Spinal analgesia
- PCA group (Active Comparator): PCA Morphine is set to the patient for 48 hours postoperative. 2 mg. of morphine is given to a patient as much as patient requires, maximum at every 7 minutes.
  Interventions: Drug: Patient Control Analgesia (PCA) Morphine

INTERVENTIONS:
Drug: Spinal analgesia — isobaric bupivacaine 0.5% 10 mg together with preservative-free morphine was injected. The dose of morphine was based on patient's age, with 200 μg in patients aged ≤ 75 years and 150 μg in patients aged > 75 years.
  Other Names: Spinal block, intrathecal block
  Arms: Spinal group
Drug: Patient Control Analgesia (PCA) Morphine — PCA Morphine is set to the patient for 48 hours postoperative. 2 mg. of morphine is given to a patient as much as patient requires, maximum at every 7 minutes.
  Other Names: Patient Control Analgesia Morphine.
  Arms: PCA group

SUMMARY:
This is a blinded randomized controlled trial in patients undergoing laparoscopic colon surgery. The aim of this study is to assess whether spinal analgesia with a mixture of bupivacaine and morphine provides better pain relief than systemic morphine in a group of patients undergoing colonic resection and using the Enhanced Recovery After Surgery (ERAS) program.

Twenty patients will receive spinal analgesia and twenty patients will receive only Patient Control Analgesia (PCA).

DETAILED DESCRIPTION:
This is a blinded randomized controlled trial in patients undergoing laparoscopic colon surgery. The aim of this study is to assess whether spinal analgesia with a mixture of bupivacaine and morphine provides better pain relief than systemic morphine in a group of patients undergoing colonic resection and using the ERAS program.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo laparoscopic colonic resection

Exclusion Criteria:

* patients who have trouble to understand, read or communicate either in French or in English
* dementia
* patients suffering from severe physical disability (arthritis, neuromuscular dysfunction, stroke, paraplegia) or inability to walk or conduct daily activity
* patients suffering from severe cardiac or respiratory disease (status ASA IV)
* patients suffering from metastatic carcinoma
* patients who have a history of chemoradiation within the six months preceding surgery
* morbid obesity
* contraindication to spinal analgesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
postoperative pain | daily during hospitalization up to 3 days after the operation

SECONDARY OUTCOMES:
opioid consumption | daily during hospitalization up to 3 days after the operation
opioid side effects | daily during hospitalization, participants will be followed for the duration of hospital stay, an expected average of 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, Professor, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada